CLINICAL TRIAL: NCT04059887
Title: Evaluation of Blood Tumor Mutation Burden (TMB) for Improved Efficacy of Atezolizumab in 2nd Line Non-small Cell Lung Cancer (NSCLC) [BUDDY]
Brief Title: Evaluation of Blood TMB for the Efficacy of Atezolizumab [BUDDY]
Acronym: BUDDY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, In-Jae, Oh, MD, Professor, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H2019-0351
Record Dates: First submitted 2019-08-09; First posted 2019-08-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lung Neoplasm Malignant
Keywords: Non-small cell lung cancer; Immune checkpoint inhibitor; Tumor mutation burden
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab (Experimental): Atezolizumab 1200 mg will be administrated every 3 week cycle
  Interventions: Drug: Atezolizumab Injection [Tecentriq]

INTERVENTIONS:
Drug: Atezolizumab Injection [Tecentriq] — Blood sampling will be performed before and after 3rd cycle of atezolizumab for evaluation of tumor mutation burden
  Other Names: Tecentriq

SUMMARY:
This is single arm, prospective, multi-center, cohort study to evaluate blood TMB for improved efficacy of atezolizumab in locally advanced or metastatic NSCLC at the study enrollment who failed one or more prior lines of chemotherapy including at least 1 platinum-based.

DETAILED DESCRIPTION:
Atezolizumab is approved as the treatment of patients with locally advanced or metastatic NSCLC who have disease progression during or following platinum-containing chemotherapy by the Ministry of Food and Drug Safety (MFDS) and the treatment is available on the National Health Insurance Service in South Korea. Patients will be treated with atezolizumab until loss of clinical benefit or unmanageable toxicity as routine practice.

In this study, the investigators will register patients who have a plan to be treated with atezolizumab as MFDS approval condition and meet study inclusion and exclusion criteria. The investigators will collect study related information during routine practice and collect blood and/or tissue(optional) samples to conduct the study.

Tumor assessment will be performed by investigator on the base of RECIST (version 1.1) and related information will be collected until disease progression for patients who have discontinued treatment. However, it will be collected until treatment discontinuation for patients who continue to receive atezolizumab following initial disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Ability to comply with protocol
3. Aged ≥ 18 years
4. Histologically or cytologically confirmed NSCLC that is locally advanced or metastatic (i.e., Stage IIIB not eligible for definitive chemoradiotherapy, Stage IV, or recurrent) NSCLC at the study enrollment
5. Disease progression during or following treatment with a prior platinum-containing regimen for NSCLC

   * Patients may have received one or more additional cytotoxic chemotherapy regimen.
   * Patients with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic tumor aberrations should have disease progression on approved therapy for these aberrations prior to receiving atezolizumab.
6. Measurable disease, as defined by RECIST v1.1 Measurable disease is defined by the presence of at least one measurable lesion by RECIST v1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
8. Life expectancy ≥ 12 weeks
9. Adequate hematologic and end organ function:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   * White blood cell (WBC) counts > 2.5 x 109/L
   * Hemoglobin ≥ 8.0 g/dL
   * Total bilirubin ≤ 2.5 X upper limit of normal (ULN) Patients with known Gilbert's disease who have serum bilirubin level ≤ 3 x ULN may be enrolled.
   * Aspartate aminotransferase (AST), alanine transaminase (ALT), and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:

Patients with documented liver metastases: AST and ALT ≤ 5 × ULN Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN

Exclusion Criteria:

1. Active or untreated central nervous system (CNS) metastases Patients with a history of treated CNS metastases that are asymptomatic are eligible
2. Malignancies other than NSCLC within 5 years prior to study enrollment, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, or ductal carcinoma in situ treated surgically with curative intent)
3. Pregnant and lactating women

   • Women of childbearing potential should use effective contraception during treatment with atezolizumab and for at least 5 months following the last dose.
4. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to study enrollment
5. Patients with autoimmune disorder or a history of chronic or recurrent autoimmune disorder

   * Patients with a history of autoimmune-mediated hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
   * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.
6. Uncontrolled idiopathic pulmonary fibrosis or drug-induced pneumonitis
7. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to study enrollment

   • Treatment with inhaled corticosteroid or megesterol acetate is permitted.
8. Patient with a known hypersensitivity to atezolizumab or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | At the end of cycle 3 (each cycle is 21 days)
  ORR between blood TMB-High vs. Low group

SECONDARY OUTCOMES:
Progression-free survival (PFS) | At the end of cycle 3 (each cycle is 21 days)
  PFS in Intention-to-treat (ITT) population and subgroups according to blood TMB and programmed cell death-1 (PDL1) status
Safety profile | Through study completion, an average of 1 year
  Incidence of Treatment-related Adverse Events as assessed by CTCAE version 4

CONTACTS AND LOCATIONS:
Overall Officials: In-Jae Oh, MD, PhD, Principal Investigator — Chonnam National Univeristy Hwasun Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim ST, Cristescu R, Bass AJ, Kim KM, Odegaard JI, Kim K, Liu XQ, Sher X, Jung H, Lee M, Lee S, Park SH, Park JO, Park YS, Lim HY, Lee H, Choi M, Talasaz A, Kang PS, Cheng J, Loboda A, Lee J, Kang WK. Comprehensive molecular characterization of clinical responses to PD-1 inhibition in metastatic gastric cancer. Nat Med. 2018 Sep;24(9):1449-1458. doi: 10.1038/s41591-018-0101-z. Epub 2018 Jul 16. PMID 30013197
- [Result] Gandara DR, Paul SM, Kowanetz M, Schleifman E, Zou W, Li Y, Rittmeyer A, Fehrenbacher L, Otto G, Malboeuf C, Lieber DS, Lipson D, Silterra J, Amler L, Riehl T, Cummings CA, Hegde PS, Sandler A, Ballinger M, Fabrizio D, Mok T, Shames DS. Blood-based tumor mutational burden as a predictor of clinical benefit in non-small-cell lung cancer patients treated with atezolizumab. Nat Med. 2018 Sep;24(9):1441-1448. doi: 10.1038/s41591-018-0134-3. Epub 2018 Aug 6. PMID 30082870